CLINICAL TRIAL: NCT05971004
Title: Effectiveness of Hydrolyzed Collagen Peptide Injection for the Treatment of Collateral Ligament Pain: A Randomized Controlled Trial
Brief Title: Effectiveness of Hydrolyzed Collagen Peptide Injection for the Treatment of Collateral Ligament Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tiss'You srl (Industry)
Responsible Party: Principal Investigator, Prof. Binh Luu Thi, Prof, Tiss'You srl
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Collagen Peptide Ligament
Record Dates: First submitted 2023-07-17; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Collateral Ligament Injury of Stifle Joint
Keywords: Collateral Ligament Pain; Knee Pain; Knee Instability; Sports Trauma; Collagen Peptide Injections; Ligament Healing
MeSH Terms: interventions — Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen Peptide Group (Experimental): The Collagen Peptide Group (31 patients) received oral pain relievers (paracetamol and anti-inflammatory NSAIDs) for 3-7 days (if the pain was severe) and one injection of collagen peptide solution (Tiss'You, Republic of San Marino) at the site of the inflamed ligament attachment point (femoral condyle).
  Interventions: Device: Arthrys (Collagen Peptide solution)
- Cortison Group (Active Comparator): The Cortison Group (31 patients) received oral painkillers (paracetamol and anti-inflammatory NSAIDs) for 3-7 days (if the pain was severe) and one injection of depo-medrol at the site of inflamed ligament attachment point (femoral condyle), combined with oral slow-acting symptomatic drugs (glucosamine 1500mg, atrodar 50mg) for 3 consecutive months.
  Interventions: Drug: Depo medrol

INTERVENTIONS:
Device: Arthrys (Collagen Peptide solution) — one injection of collagen peptide solution (Tiss'You, Republic of San Marino) at the site of the inflamed ligament attachment point
  Arms: Collagen Peptide Group
Drug: Depo medrol — one injection of depo-medrol at the site of inflamed ligament attachment point (femoral condyle), combined with oral slow-acting symptomatic drugs (glucosamine 1500mg, atrodar 50mg) for 3 consecutive months.
  Arms: Cortison Group

SUMMARY:
Conducted by Binh Luu Thi, Lan Tran Thi, and Minh Hang Hoang Thi at Thai Nguyen National Hospital, the study investigates a new approach to treating persistent collateral ligament pain, common among athletes. The research examines the therapeutic use of hydrolyzed collagen peptide injections, a treatment that addresses pain and inflammation in ways previous methods have not.

The study involves a randomized controlled trial with 62 patients, all diagnosed with inflammation in the collateral ligament site. The patients are split into two groups: one receiving collagen injections alongside oral painkillers and the other receiving depo-medrol injections with oral painkillers.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years,
* lateral knee pain with a duration of 3 months or longer,
* ultrasound evidence of inflammation of the femoral condyle attachment point,
* agreement to participate in the study

Exclusion Criteria:

* trauma,
* infection,
* dermatitis at the site of the inflammation,
* damage to surrounding knee structures,
* history of chronic inflammatory arthritis (such as gout or rheumatoid arthritis),
* local corticosteroid injection within 3 months before participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
WOMAC | 6 months
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) assessing functionality from 0 to 96 for the total WOMAC where 0 represents the best health status and 96 the worst possible status.

SECONDARY OUTCOMES:
VAS (Visual Analogue Pain) | Baseline, 3 months, 6 months
  Visual Analogue Pain assessing pain from 0 (no pain) to 10 (unbearable pain)
Ultrasound | Baseline, 3 months, 6 months
  Ultrasound evaluation for hypoechoic (signal reduction), normal, and hyperechoic (signal amplification) ligaments. Hypoechoic signal suggests damage or degeneration of the ligament; normal signal suggests healthy ligament tissue; hyperechoic signal suggests calcification, scar, or inflammation.
Likert | Baseline, 6 months
  Likert scale for patients' satisfaction from 1 (no statisfaction) to 5 (maximum satisfaction)
WOMAC | Baseline, 3 months
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) assessing functionality from 0 to 96 for the total WOMAC where 0 represents the best health status and 96 the worst possible status.

CONTACTS AND LOCATIONS:
Locations (1):
- Tiss'You, Domagnano, RSM, San Marino

IPD SHARING:
Plan to Share IPD: No